CLINICAL TRIAL: NCT01865903
Title: Nutritional Problems and Changes in Body Composition in Patients With Non-small Cell Lung Cancer; Incidence, Development and Impact on Quality of Life, Adverse Effects and Survival.
Brief Title: Nutritional Problems and Changes in Body Composition in Patients With Non-small Cell Lung Cancer (LEKS)
Acronym: LEKS
Status: Terminated | Type: Observational
Why Stopped: To Low recruitment and competing studies
Sponsor: Oslo University Hospital (Other)
Collaborators: Diakonhjemmet Hospital (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Kjersti Hornslien, MD, Oslo University Hospital
Other Study IDs: 2012/830/REK sør-øst D
Record Dates: First submitted 2013-05-08; First posted 2013-05-31 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Weight Loss; Cachexia
Keywords: NSCLC; sarcopenia; cachexia
MeSH Terms: conditions — Weight Loss; Cachexia; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsamples for biobank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: All with diagnose of NSCLC in Oslo during 6 months
- Cohort 2: All NSCLC in Ulleval university hospital whom are in need of palliative chemotherapy

SUMMARY:
Weight loss and loss of lean body mass are common and associated with adverse outcomes such as loss of strength, reduced immune- and pulmonary function and increased disability in advanced cancer. Progressive weight loss interferes with cancer therapy and is responsible for reduced quality of life (QoL) as well as shorter survival irrespective of tumour mass or presence of metastases. Weight loss in advanced cancer is regarded as a major clinical challenge because of its serious consequences, its varying aetiology and the contribution of multiple pathophysiological mechanisms that are poorly disentangled.

DETAILED DESCRIPTION:
Weight loss and loss of lean body mass are common and associated with adverse outcomes such as loss of strength, reduced immune- and pulmonary function and increased disability in advanced cancer. Progressive weight loss interferes with cancer therapy and is responsible for reduced quality of life (QoL) as well as shorter survival irrespective of tumour mass or presence of metastases. Weight loss in advanced cancer is regarded as a major clinical challenge because of its serious consequences, its varying aetiology and the contribution of multiple pathophysiological mechanisms that are poorly disentangled.

The main contributor to weight loss in advanced cancer is considered to be development of cancer cachexia. The term refers to a syndrome of progressive loss of body weight and muscle atrophy involving two parallel pathways, i.e. negative energy balance and inflammation-driven catabolism. The negative energy balance may be a direct result of malnutrition caused by cancer and treatment related symptoms that interfere with food intake and routine assessment of nutritional status is therefore advocated. The interaction and relative contribution of these pathways in the development of cancer cachexia are, however, poorly understood. Through novel use of traditional clinical data and biological markers, we propose to investigate the interplay and magnitude of the processes involved in the development of cancer cachexia. This will contribute to a new understanding that may lead to more precise identification of remediable factors and improved treatment. In this context, we will also investigate the relevance of using screening tools for nutritional status, as advocated by the Norwegian Health Authorities. However, in advanced cancer the identifying ability of the recommended screening tools is poorly documented.

The present study is part of a larger project by our group. The overall project includes two parallel studies based on the same comprehensive data collection, targeting patients with non-small cell lung cancer (NSCLC). Tumours of the lung are one of the most common causes of cancer related weight loss. These patients are therefore an ideal target for studying the mechanisms and impact of nutritional problems and cachexia, as proposed in the present study. The other parallel study, which is approved by the Regional Committee for Medical and Health Research Ethics (REC), Region South East (2012/830), aims at describing the frequency and development of weight loss in NSCLC patients, and its relation to tumour stage, response and side effects of chemotherapy.

This study also makes part of a larger research effort focusing on cachexia and changes in body composition in cancer patients by our group. A study on the impact of sarcopenia (severe muscle loss) in NSCLC is ongoing as well a prospective study on cachexia in pancreatic cancer, using the same assessments as the present study. The present study will significantly contribute to the understanding of the mechanisms of weight loss and cachexia in advanced cancer in general and in NSCLC in particular, and will provide knowledge that is needed to improve medical treatment and follow-up of a large group of patients. Thus, the study is in line with the research strategy from the South-Eastern Norway Regional Health Authority (South-Eastern Norway RHA). Furthermore, the study emerges from a multidisciplinary research network representing several areas of medical and nutritional expertise and with an established international partnership.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NSCLC.
* No other active cancer.
* Must be able to consent.
* Fluent in Norwegian.

Exclusion Criteria:

* Other active cancer than NSCLC
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 250 new cases of lung cancer are diagnosed in Oslo every year. About 200 of these belong to the defined catchment area for the present study. Approximately 150 patients are expected to be in a palliative setting. Based on the number of new referrals to OUS Ullevål in 2011, about 60-80 patients with NSCLC will be starting first line palliative chemotherapy every year. A sample size of 110 patients is planned for this study Cohort 2, which gives an enrolment period of about 2 years In Cohort 1 another 50 patients.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-06-15 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Nutritional Problems and Changes in Body Composition in Patients With Non-small Cell Lung Cancer (LEKS) | 30months
  To describe the status of nutrition and body composition in all patients with non small cell lung cancer at the moment of diagnose in a certain period of time, and to follow the possible changes in the same in those patients who then afterwards receive palliative chemotherapy.

SECONDARY OUTCOMES:
The relation between nutrition, tumor burden and outcome | 30 months
  1. The interaction between negative energy balance and inflammation-driven catabolism, and tumor burden and analyse the predictive impact on QoL and survival

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway